CLINICAL TRIAL: NCT00180960
Title: Treatment of a Cancerous Disease of the Peritoneum With Complete Cytoreductive Surgery With Intraperitoneal Chemohyperthermia Using Oxaliplatin Plus Irinotecan
Brief Title: Treatment of a Cancerous Disease of the Peritoneum With Complete Cytoreductive Surgery and Intraperitoneal Chemohyperthermia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHIP4 Phase II
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Colon Tumors; Rectum Tumors; Appendix Tumors; Peritoneum Tumors; Endocrine Tumors
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Appendiceal Neoplasms | interventions — Oxaliplatin; Irinotecan

INTERVENTIONS:
Drug: Oxaliplatin and irinotecan

SUMMARY:
The purpose of this study is to evaluate the treatment of a cancerous disease of the peritoneum with complete cytoreductive surgery with intraperitoneal chemohyperthermia using oxaliplatin plus irinotecan.

This is a Phase II study with 100 patients. Origins of the tumors: these include colon, rectum, appendix, peritoneum, and endocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal seedings coming from colon, rectum, pseudomyxoma (appendix), peritoneum (mesothelioma and serous tumors), or endocrine tumors.
* No extra-abdominal metastases
* Good general status (American Society of Anesthesiologists Physical Status score [ASA] 1 or 2)
* Signed consent

Exclusion Criteria:

* Tumor seedings coming from other origins
* Huge peritoneal carcinomatosis (peritoneal score > 25, except for pseudomyxomas)
* Peritoneal carcinomatosis progressing rapidly
* Presence of extra-abdominal metastases
* Patients presenting contraindications to the use of oxaliplatin or irinotecan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-06

PRIMARY OUTCOMES:
To study overall survival

SECONDARY OUTCOMES:
To study mortality-morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Elias, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave-Roussy, Villejuif, France